CLINICAL TRIAL: NCT01848717
Title: A Single-Center, Single Arm, Pre-post Test Design, Open Clinical Study to Evaluate the Efficacy and Safety of MINTLIFT® Group for Nasolabial Fold
Brief Title: Evaluate the Efficacy and Safety of MINTLIFT® Group for Nasolabial Fold
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: HansBiomed Co.,Ltd. (Industry)
Responsible Party: Principal Investigator, Beom Joon Kim, Associate Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HANS_MINTLIFT_1101
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Nasolabial Fold

ARMS (1):
- Lift thread (Experimental)
  Interventions: Device: MINTLIFT®

INTERVENTIONS:
Device: MINTLIFT®

SUMMARY:
The objective of this clinical test is to verify the safety and efficacy of MINTLIFT®, used for the purpose of improving the appearance of the nasolabial fold on both sides of the face.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who desire an improvement in the appearance of the nasolabial fold on both sides of the face and who have a score of 3 or 4 on the Wrinkle Severity Rating Scale (WSRS) at the time of the screening and at the baseline time point
* Individuals who have consented to abstain from any other dermatological procedures or treatments, including treatments for wrinkle reduction in the facial area, during the duration of this clinical test

Exclusion Criteria:

* Subjects who have a scar or hypertrophic scar or a history of keloid conditions that may affect the determination of effect
* Subjects allergic to local anesthetics or sleep anesthetics
* Subjects whose ALT/AST ratio is 2.5 times or more greater than the normal upper limit
* Subjects who have been administered an anticoagulant (with the exception of low dosage aspirin (100mg, up to 300mg/day)) within 2 weeks of the date of the screening, or who require an anticoagulant during the period of the clinical test
* Subjects who have been administered systemic corticosteroids or anabolic steroids within two weeks of the date of the screening or who require their administration during the period of the clinical test (note, however, that the administration of inhaled corticosteroids in a standardized dosage is permissible)
* Subjects who have been administered Vitamin E or non-steroidal anti-inflammatory drugs within 1 week of the date of the screening
* Subjects who have used Topical liniments in the facial area (steroids, retinoids: only medical drugs are included in this criteria, with the exclusion of cosmetic products) within 4 weeks of the date of the screening or who plan on continuing usage during the period of the clinical test
* Subjects who have received wrinkle reduction treatment using CaHA within 1 year of the date of the screening
* Subjects who have received wrinkle reduction treatment using collagen or HA filler within 6 months of the date of the screening, or who have received acne treatment, skin regeneration procedures, or cosmetic surgical procedures (including Botox injections) in the facial area
* Subjects who have a permanent skin expanding implant such as Softform or silicon inserted in the facial area
* Subjects who have scars in the facial area requiring treatment that has not healed for a period of 1 year or longer, or who have a scar or trace in the area on which the clinical test device will applied.
* Subjects who have a chronic or recurrent infection or a history of inflammatory disease that may affect this clinical test
* Subjects who have experienced severe allergies such as symptoms of anaphylaxis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of the subjects who demonstrated wrinkle improvement to -1 or below in WSRS as determined by an independent evaluator | 12th week of the application of the test device
  The percentage of the subjects within the test group who demonstrated wrinkle improvement to -1 or below in WSRS in the 12th week following the application of the device in comparison to the condition prior to the application (12th week- prior to application) as determined by an independent evaluator

SECONDARY OUTCOMES:
The percentage of the subjects who demonstrated wrinkle improvement to -1 or below in WSRS as determined by an independent evaluator | in the 4th, 8th and 24th week following the application of the device
The percentage of the subjects who demonstrated wrinkle improvement to -1 or below in WSRS as determined by the investigator | in the 4th, 8th, 12th and 24th week following the application of the device
The average of the differences between the baseline and the WSRS evaluated by the independent evaluator | in the 4th, 8th, 12th and 24th week following the application of the test device
The average of the differences between the baseline and the WSRS evaluated by the subject | in the 4th, 8th, 12th and 24th week following the application of the test device
The average value of Global Aesthetic Improvement Scale (GAIS) scores as determined by the investigator and the distribution of scores | in the 12th and 24th week following the application of the test device
The average value of GAIS scores as determined by the subject and the distribution of scores | in the 12th and 24th week following the application of the test device

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon KIM, MD, PhD, Principal Investigator — Department of Dermatology
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea